CLINICAL TRIAL: NCT05665231
Title: Morphometric, Imaging and Photographic Comparison of Peri-implant Tissues Between V3 and C1 Mis ® Implants in Post-extraction Alveolus in the Anterior Region of the Maxilla
Brief Title: Differences Between Two Type Implants in Post-extraction Alveolus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 080237
Record Dates: First submitted 2022-11-04; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-10

CONDITIONS: Dental Implants, Single-Tooth
Keywords: dental implants; extraction socket; immediate placement; implant geometry
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Intervention Model Description: The sample consists of 20 clinical cases of unitary tooth loss in the region of the incisors, canines, and maxillary premolars of patients from the clinic of the Faculty of Dental Medicine of the University of Porto. Clinical cases were randomly grouped into 2 implant groups (triangular shape - implant V3 form Mis® and cylindrical shape - implant C1 from Mis®) by a closed envelope allocation (triangular shape implant: 10 clinical cases; cylindrical shape: 10 clinical cases). Three consecutive measurements were performed for each parameter, using their average for statistical analysis. The envelopes were prepared prior to the start of the clinical study, mixed and stored. before each surgery, an envelope was randomly taken for the preparation of the surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The envelopes were prepared prior to the start of the clinical study, mixed and stored. before each surgery, an envelope was randomly taken for the preparation of the surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V3 Mis® implant (Experimental): Implant with coronal triangular neck
  Interventions: Other: A - Bone defect (clinical variables); Other: B- Bacterial plaque index (O'Leary index)(clinical variables); Other: C- Probing depth; Other: D- Bleeding on probing; Other: E- Gingival phenotype; Other: F- Implant insertion torque (Clinical variables); Other: G- Implant stabilization quotient (ISQ) (clinical variables); Other: Morphometric results (Direct measurements - millimeter); Other: Morphometric results (plaster models measurements - millimeter); Other: Imaging Results (X-ray) (millimeter); Other: Imaging Results (CBCT)(millimeter); Other: Photographic results PES/WES index
- C1 MIS® implant (Active Comparator): Implant with coronal cylindrical neck (regular)
  Interventions: Other: A - Bone defect (clinical variables); Other: B- Bacterial plaque index (O'Leary index)(clinical variables); Other: C- Probing depth; Other: D- Bleeding on probing; Other: E- Gingival phenotype; Other: F- Implant insertion torque (Clinical variables); Other: G- Implant stabilization quotient (ISQ) (clinical variables); Other: Morphometric results (Direct measurements - millimeter); Other: Morphometric results (plaster models measurements - millimeter); Other: Imaging Results (X-ray) (millimeter); Other: Imaging Results (CBCT)(millimeter); Other: Photographic results PES/WES index

INTERVENTIONS:
Other: A - Bone defect (clinical variables) — At T0, the edentulous space to be rehabilitated will be characterized in terms of the morphometric level of the existing defect in the vestibular cortical, according to the classification by Caplanis N. in EDS-1 or EDS-2.
Other: B- Bacterial plaque index (O'Leary index)(clinical variables) — At time T-1 and T4, the investigator will analyse the existing plaque on teeth adjacent to the surgical site using a dichotomous score (0 = no visible plaque at the soft tissue margin, 1 = visible plaque at the soft tissue margin). The result will be present in percentage (0% (better)-100%(worse)) and will describe the change between T-1 and T4, and compare the results between implants type.
Other: C- Probing depth — At Time T-1 and T4, the investigators will analyse the probing depth of the teeth adjacent to the site to be treated at 6 points: mesiobuccal, vestibular, distobuccal, mesiopalatal, palatine, distopalatal. The recordings will be carried out with a CP 15 UNC, Hu-Friedy® Chicago, IL, EUA manual probe.The result will be present in millimeters. The change between T-1 and T4 is also going to be analysed and compare implants results.
Other: D- Bleeding on probing — At time T-1 and T4, the investigators will analyse the bleeding on probing of the teeth adjacent to the site to be treated at 6 points: mesiobuccal, vestibular, distobuccal, mesiopalatal, palatine, distopalatal. The recordings of bleeding on probing will be carried out with a CP 15 UNC, Hu-Friedy® Chicago, IL, EUA manual probe.The result will be present in percentage (0% (better)-100%(worse)) and will describe the change between T-1 and T4 and compare between implants type.
Other: E- Gingival phenotype — At time T-1, the identification of the gingival phenotype is performed by clinical inspection with a periodontal probe. The gingival phenotype will be classified as thin, moderate or thick. The investigators will compare implant results.
Other: F- Implant insertion torque (Clinical variables) — Recording of implant insertion torque, in Ncm during placement in T1, and compare implants results.
Other: G- Implant stabilization quotient (ISQ) (clinical variables) — Determination of the implant stability coefficient at the time of implant placement (T1) and in the 2nd surgical phase (T3) using the Osstell® device (minimum 1; maximum 100; high stability when ≥70) and analysis of the change between T1 and T3 and different implants results.
Other: Morphometric results (Direct measurements - millimeter) — Compare Direct measurements (millimeters) at the different times intervention with periodontal probe or gauge and analyse the change between times and compare implant results.
  In T-1, T2 and T3c and T4 the investigators will evaluate interdental distance; BPD, cortical bone, papilla and volume, corresponding of measurements: a,b,c and r.
  In T0, the investigators will evaluate interdental distance; BPD, cortical, bone and global volume corresponding to measurements: a, b, c, d, e, q, r, s, t, and u).
  In T1 e T3, the investigators will evaluate interdental distance; BPD, cortical, bone and global volume, implant parameter corresponding to measurements: a, b, d, e, f, g, h, I, j, k, l, m, n, p, q, r and ISQ value.
Other: Morphometric results (plaster models measurements - millimeter) — Preparation of plaster models at times T-1 and T4 and the following measurements (millimeter) will be evaluated with the use of periodontal probe or gauge and will analyse the change between T-1 and T4 and compare implants results:
  1. interdental distance
  2. bucco-palatal distance (BPD)
  3. presence of papilla
  r. global volume.
Other: Imaging Results (X-ray) (millimeter) — The investigator will measure (millimeters, using the imaging software virtual ruler) the results of digital X-ray at times T-1, T1,T4 and analyse the variation and compare implants results. The measurements are:
  a. interdental distance; i. implant - cemento-enamel junction (CEJ) of adject teeth distance; l. distance from the implant position depth to the buccal bone crest; n. implant diameter; o. implant length.
Other: Imaging Results (CBCT)(millimeter) — The investigator will measure (millimeters, using the imaging software virtual ruler) the results of CBCT at times T-1 and T4, analyse the variation and compare implants results. The measurements are:
  1. interdental distance;
  2. bucco-palatal distance (BPD);
  d. buccal cortical distance; e. palatal cortical distance; f. mesial cortical distance; g. distal cortical distance; h. jumping distance; j. buccal cortical wall-implant distance; k. jumping distance space depth; l. distance from the implant position depth to the buccal bone crest; m. distance from the buccal cortex to the center of the implant; n. implant diameter; o. Implant length; q. global bone volume; r. global volume; s. alveolus buccal-palatal distance; t. alveolus mesial-distal distance; u. alveolus depth.
Other: Photographic results PES/WES index — The investigator will analyse the intraoral photographs to describe the Pes/Wes index, in time T-1 (initial) and T4 (final), and compare the PES/WES results between implants.The score will range on 0-10, the best score is ≥8.

SUMMARY:
One of the challenges of current implantology involves the preservation or reduction of existing bone resorption, mainly in the buccal bone plate, after tooth loss, which becomes of special importance in the anterior region of the maxilla (aesthetic region). The study evaluates the macroscopic shape of neck implant influence in the results of immediate implants, in a population comprised of individuals from the clinic of the Faculty of Dental Medicine of the University of Porto in need of replacement of a single tooth. It is intended to evaluate the morphometric (direct measures and plaster models measurements), imaging, and photographic characteristics of the V3 implant in comparison with the C1 implant of Mis® by an evaluation period of 6 months when placing an immediate implant.

DETAILED DESCRIPTION:
The study is a prospective randomized clinical trial performed by a single investigator, without a control group. The project was designed in 2016 and the participants were recruited between 2017 and 2021.

Patients who met the inclusion criteria were recruited by the Unit of Oral Surgery and Implantology of the University of Porto from 2017 to 2021. The patients were fully informed of the characteristics of the study and were invited to participate. A complete medical history was taken for each of the patients, and they also underwent a thorough oral examination. The investigation was carried out in accordance with the criteria recommended in the CONSORT Guidelines.

1. Sample characterization The sample will consist of clinical cases of unitary tooth loss in the region of incisors, canines, and maxillary premolars of patients from the clinic of the Faculty of Dental Medicine of the University of Porto. The study follows ethical principles of the Ethics Committee of the Faculty of Dental Medicine, University of Porto, and guidelines from the Declaration of Helsinki for clinical trials with humans.

   Thus, after informed consent, the patients will be randomly grouped into 2 groups, through a closed letter draw:

   Group I- patients submitted to the protocol of immediate placement of the V3 Mis® implant; Group II- patients submitted to the protocol of immediate placement of C1 MIS® implant.
2. Surgical protocol

   Surgical protocol for implant placement (1st surgical phase):

   Starting with a local anesthetic administration, the incision and elevation of the mucoperiosteal flap are performed. Then the tooth is atraumatically extracted with odontosection and use of mucoperiosteal elevators, and the socket is cleaned with saline solution. After this is complete, the osteotomy for implant placement is performed, and the implant and the healing cap are placed. Finally, the implant is submerged and the surgical wound is sutured with non-resorbable 4/0 polyamide thread. For the provisional a Maryland crown was performed. Individuals are monitored monthly during the healing phase, and sutures are removed after 7 days.

   Pre- and post-operative therapy includes:
   * Antibiotic: amoxicillin, 1g (twice a day for 8 days), and in case of allergy, clarithromycin 500mg (twice a day for 8 days). Administration started on the day of surgery;
   * Anti-inflammatories (diclofenac 50mg, twice a day, for 4 to 5 days);
   * Chlorhexidine (0.2%) rinses (twice a day for 21 days).

   Surgical protocol for placement of a healing abutment (2nd surgical phase):

   Starting with a local anesthetic administration, the incision and elevation of the mucoperiosteal flap are performed. After, the healing screw is removed and the implant healing abutment (with 3x5,8mm) is placed. Finally, the surgical wound is sutured with non-resorbable 4/0 polyamide thread. Suture removal is performed after 7 days. After healing, impressions were made for the fabrication of a screw-retained cad-cam crown with platform switching concept.

   The investigators chose open flap implant placement without bone or connective graft placement, or immediate provisional, and direct measurement of hard and soft tissues to study the differences between implants. The goal is to evaluate only the effect of the type of coronal shape implant, minimizing the influence of other factors that could lead to bias errors.
3. Evaluations over time

T-1 - First visit pre-operative:, Morphometric evaluation (clinical direct measurements and plaster models measurements), imaging (X-ray and CBCT) and photographic (PES/WES) analysis.

T0 - Extraction tooth: Morphometric (clinical direct measurements) and imaging (X-ray) evaluation.

T1 - Implant placed (1st surgical phase): Morphometric (clinical direct measurements) and imaging evaluation (X-ray) evaluation.

T2 - 2 months submerged: Morphometric evaluation (clinical direct measurements).

T3 - Healing abutment (2nd surgical phase - 4 months): Morphometric evaluation (clinical direct measurements).

T3c - Definitive Crown: Morphometric evaluation(clinical direct measurements).

T4 - 6 months osteointegration: Morphometric evaluation (clinical direct measurements and plaster models measurements), imaging (X-ray and CBCT) and photographic (PES/WES) analysis.

4 - Observed clinical variables:

A- Bone defect: the edentulous space to be rehabilitated will be characterized in terms of the morphometric level of the existing defect in the vestibular cortical, according to the classification by Caplanis N., at time T0, in EDS-1 or EDS-2.

B- Bacterial plaque index (O'Leary index): an analysis will be performed for existing plaque on teeth adjacent to the surgical site using a dichotomous score (0 = no visible plaque at the soft tissue margin, 1 = visible plaque at the soft tissue margin).

C- Probing depth: analysis of the probing depth of the teeth adjacent to the site to be treated at 6 points: mesiobuccal, vestibular, distobuccal, mesiopalatal, palatine, distopalatal. The recordings will be carried out with a CP 15 UNC, Hu-Friedy® Chicago, IL, EUA manual probe.

D- Bleeding on probing: performed at the 6 locations around adjacent teeth when analyzing the probing depth.

E- Gingival phenotype: identified by clinical inspection with a periodontal probe.

F- Implant insertion torque: recording of implant insertion torque during placement (T1).

G- Implant stabilization quotient (ISQ): determination of the implant stability coefficient at the time of implant placement (T1) and in the 2nd surgical phase (T3) using the Osstell® device, the resonance frequency analysis is performed.

5 - Morphometric analysis

Measurements to be assessed:

1. interdental distance: distance measured using the straight gauge between adjacent teeth at the bone crest.
2. bucco-palatal distance (BPD): distance measured by the thickness gauge in the midline of the edentulous space between the buccal edge of the buccal cortex to the palatal edge of the palatal cortex.
3. presence of papilla: evaluation through the pink aesthetics index (Pink Esthetic Score - PES, proposed by Fürhauser and collaborators, white aesthetics index (White Esthetic Score - WES, proposed by Belser UC).
4. buccal cortical distance: thickness of the buccal cortical through the thickness gauge, measured at the midline of the alveolus.
5. palatal cortical distance: thickness of the palatal cortical through the thickness gauge, measured at the midline of the alveolus.
6. mesial cortical distance: thickness of the palatal cortical through the thickness gauge, measured at the midline of the alveolus.
7. distal cortical distance: thickness of the palatal cortical through the thickness gauge, measured at the midline of the alveolus.
8. jumping distance: distance between the inner of the buccal or palatal or mesial or distal cortex and the buccal surface of the implant measured using the periodontal probe;
9. implant - cemento-enamel junction (CEJ) of adject teeth distance: determination of the vertical dimension from the occlusal surface of the implant to the cemento-enamel junction of adjacent teeth with a periodontal probe, in mesial and distal sides.
10. buccal cortical wall-implant distance: using the periodontal probe, horizontal dimension between the buccal surface of the cortical and the buccal surface of the implant, at buccal, palatal, mesial and distal cortical.
11. jumping distance space depth: maximum depth of the space between the buccal cortex and the implant wall through the periodontal probe at buccal, palatal, mesial and distal cortical.
12. distance from the implant position depth to the buccal bone crest: vertical dimension of the occlusal surface of the implant in relation to the bone crest through the periodontal probe, at buccal, palatal, mesial and distal cortical.
13. distance from the buccal cortex to the center of the implant: horizontal dimension from the buccal edge of the buccal cortex to the center of the implant with a periodontal probe, at buccal, palatal, mesial and distal cortical.
14. implant diameter: diameter of the implant.
15. Implant length: length of the implant.
16. soft tissue thickness: Soft tissue thickness was assessed using the thickness gauge at the buccal and palatal mucosa.
17. global bone volume: using the periodontal probe and thickness gauge, horizontal dimension between the buccal surface of the buccal cortical and the lingual surface of the palatal cortical, at the bone crest and 3 mm below this.
18. global volume: Soft and hard tissue thickness was assessed using the periodontal probe and thickness gauge, at the crest and 3 mm below this.
19. alveolus buccal-palatal distance: with periodontal probe.
20. alveolus mesa-distal distance: with periodontal probe.
21. alveolus depth: with periodontal probe.

    The morphometric analysis will be performed in all patients as follows:

    5.1- Clinical direct measurements in mouth:

    Direct measurements will be carried out using a thickness gauge and periodontal probe ( CP 15 UNC, Hu-Friedy® Chicago, IL, EUA manual probe), with a 0.5mm. The appropriate measures will be applied, according to the chronograms times.

    5.2- Plaster models measurements: Initial impressions will be made at time T-1 to prepare a thermoformed gutter with calibration traces for measurements at different surgical times.

    Preparation of plaster models at times T-1 and T4 and different measurements will be evaluated.

    6 - Imaging analysis

    6.1- Periapical X-ray: Use of the parallelism technique and use of thermoformed gutter with horizontal and vertical plane marking. Periapical x-rays will be performed at times T-1, T1,T4.

    6.2- Cone Beam Computerized Tomography (CBCT): In the analysis of maxillary computed tomography, at times T-1 and T4, with radiographic guide.

    7- Photographic analysis:

    Photographs will be taken using a Canon 450D device, a Canon Macro Lens EF 100mm lens and a Macro Ring Lite MR-14EX circular flash, with an image ratio of 1:1.

    7.1- Extra-oral photographs: Initial (T-1) and final (T4) extraoral photographs will be taken at a distance of 2.5 m for replication and with reference to the occlusal plane. The reference will be the midsagittal plane and the Frankfurt plane, and the frontal photograph will be taken in the resting and smiling position, along with a profile photograph of the patient at rest and smiling.

    7.2- Intra-oral photographs: Intraoral photographs will be taken during the treatment phases T-1 and T4 measuring a distance of 40 cm for replication and with reference to the occlusal plane. For this, lip retractors, intraoral mirrors, and black backgrounds will be used. Frontal photography in maximum occlusion, left and right lateral photography with only two adjacent teeth, and upper and lower occlusal photography will be performed.

    Evaluated measurements:

    The presence of papilla; The PES and WES index was evaluated through the analysis of photographs.

    8- Statistical analysis

    The sample size was calculated from G*Power 3.1.9.6 considering F tests - ANOVA with Repeated measures, moderate effect size (f=0.30), α= 0.05, Power (1-β err prob)=0.95 and 2 groups of implants evaluated in 7 times.

    A descriptive analysis will be presented to characterize the qualitative and quantitative variables (gender, race, and age) presented in the form of graphs and summary tables. The statistical techniques to be adopted will be in accordance with the nature of the variables under study.

    Therefore, for the evaluation of quantitative measures in time, the analysis will be proposed through the ANOVA test with repeated measures with one factor (type of implant), after verifying the conditions of normality and sphericity of the variables. Measurement error control (collection of three measurements in each observation) and examiner calibration (intra-operator variability).

    For processing the results, the IBM Statistics software version 24.0 will be used. The decision rule will be for a statistical significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Patients with understanding and free decision-making for informed consent
* Patients who need rehabilitation of a tooth in the region of incisors, canines, or maxillary premolars
* Patients with EDS-1 or EDS-2 dental sockets, according to Caplanis N. classification.

Exclusion Criteria:

* Patients with systemic pathologies that contraindicate the surgical procedure;
* Prolonged Non-steroidal anti-inflammatory drugs (NSAIDs);
* Bisphosphonate therapy;
* Lack of opposing teeth on implant site;
* Lack of adjacent teeth on implant site;
* Dental-sockets with total loss of one of the cortical;
* Untreated periodontal pathology;
* Pathology or circumstance that prevents patients from attending routine check-ups;
* Patients who smoke more than 10 cigarettes/day. Smokers are advised to reduce or stop smoking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
A - Bone defect (clinical variables) | T0
  At T0, the edentulous space to be rehabilitated will be characterized in terms of the morphometric level of the existing defect in the vestibular cortical, according to the classification by Caplanis N. in EDS-1 or EDS-2.
B- Bacterial plaque index (O'Leary index)(clinical variables) | 6 months
  At time T-1 and T4, the investigator will analyse the existing plaque on teeth adjacent to the surgical site using a dichotomous score (0 = no visible plaque at the soft tissue margin, 1 = visible plaque at the soft tissue margin). The result will be present in percentage (0% (better)-100%(worse)) and will describe the change between T-1 and T4, and compare the results between implants type.
C- Probing depth (clinical variables) | 6 months
  At Time T-1 and T4, the investigators will analyse the probing depth of the teeth adjacent to the site to be treated at 6 points: mesiobuccal, vestibular, distobuccal, mesiopalatal, palatine, distopalatal. The recordings will be carried out with a CP 15 UNC, Hu-Friedy® Chicago, IL, EUA manual probe.The result will be present in millimeters. The change between T-1 and T4 is also going to be analysed and compare implants results.
D- Bleeding on probing (clinical variables) | 6 months
  At time T-1 and T4, the investigators will analyse the bleeding on probing of the teeth adjacent to the site to be treated at 6 points: mesiobuccal, vestibular, distobuccal, mesiopalatal, palatine, distopalatal. The recordings of bleeding on probing will be carried out with a CP 15 UNC, Hu-Friedy® Chicago, IL, EUA manual probe.The result will be present in percentage (0% (better)-100%(worse)) and will describe the change between T-1 and T4 and compare between implants type.
E- Gingival phenotype (clinical variables) | T-1
  At time T-1, the identification of the gingival phenotype is performed by clinical inspection with a periodontal probe. The gingival phenotype will be classified as thin, moderate or thick. The investigators will compare implant results.
F- Implant insertion torque (Clinical variables) | T1
  Recording of implant insertion torque, in Ncm during placement in T1, and compare implants results.
G- Implant stabilization quotient (ISQ) (clinical variables) | 6 months
  Determination of the implant stability coefficient at the time of implant placement (T1) and in the 2nd surgical phase (T3) using the Osstell® device (minimum 1; maximum 100; high stability when ≥70) and analysis of the change between T1 and T3 and different implants results.
Morphometric evaluation (clinical direct measurements) | 6 months
  Compare Direct measurements (millimeters) at the different times intervention with periodontal probe or gauge and analyse the change between times and compare implant results.
  In T-1, T2 and T3c and T4 the investigators will evaluate interdental distance; BPD, cortical bone, papilla and volume, corresponding of measurements: a,b,c and r.
  In T0, the investigators will evaluate interdental distance; BPD, cortical, bone and global volume corresponding to measurements: a, b, c, d, e, q, r, s, t, and u).
  In T1 e T3, the investigators will evaluate interdental distance; BPD, cortical, bone and global volume, implant parameter corresponding to measurements: a, b, d, e, f, g, h, I, j, k, l, m, n, p, q, r and ISQ value.
Morphometric evaluation (plaster models measurements) | 6 months
  Preparation of plaster models at times T-1 and T4 and the following measurements (millimeter) will be evaluated with the use of periodontal probe or gauge and will analyse the change between T-1 and T4 and compare implants results:
  1. interdental distance
  2. bucco-palatal distance (BPD)
  3. presence of papilla
  r. global volume.
Imaging periapical X-ray evaluation (millimeter) | 6 months
  The investigator will measure (millimeters, using the imaging software virtual ruler) the results of digital X-ray at times T-1, T1,T4 and analyse the variation and compare implants results. The measurements are:
  a. interdental distance; i. implant - cemento-enamel junction (CEJ) of adject teeth distance; l. distance from the implant position depth to the buccal bone crest; n. implant diameter; o. implant length.
Cone Beam Tomography (CBCT) evaluation (millimeter) | 6 months
  The investigator will measure (millimeters, using the imaging software virtual ruler) the results of CBCT at times T-1 and T4, analyse the variation and compare implants results. The measurements are:
  1. interdental distance;
  2. bucco-palatal distance (BPD);
  d. buccal cortical distance; e. palatal cortical distance; f. mesial cortical distance; g. distal cortical distance; h. jumping distance; j. buccal cortical wall-implant distance; k. jumping distance space depth; l. distance from the implant position depth to the buccal bone crest; m. distance from the buccal cortex to the center of the implant; n. implant diameter; o. Implant length; q. global bone volume; r. global volume; s. alveolus buccal-palatal distance; t. alveolus mesial-distal distance; u. alveolus depth.
PES/WES index - Photography results | 6 months
  The investigator will analyse the intraoral photographs to describe the Pes/Wes index, in time T-1 (initial) and T4 (final), and compare the PES/WES results between implants.The score will range on 0-10, the best score is ≥8.

SECONDARY OUTCOMES:
Osseointegration survival rate | 6 months
  At the surgical second phase, it will observe the percentage of dental implant osseointegration in each group at time T4.
Biological complication | 6 months
  It will indicate and describe biological complication if they occur, at time T4.
Prosthetic complication | 6 months
  It will indicate and describe the prosthetic complication if they occur, at time T4.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Faria Almeida, PhD, Study Director — Faculdade de Medicina Dentaria da Universidade do Porto
Locations (1):
- Faculty of Dental Medicine, Porto University, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buser D, Chappuis V, Belser UC, Chen S. Implant placement post extraction in esthetic single tooth sites: when immediate, when early, when late? Periodontol 2000. 2017 Feb;73(1):84-102. doi: 10.1111/prd.12170. PMID 28000278
- [Result] Araujo MG, Sukekava F, Wennstrom JL, Lindhe J. Tissue modeling following implant placement in fresh extraction sockets. Clin Oral Implants Res. 2006 Dec;17(6):615-24. doi: 10.1111/j.1600-0501.2006.01317.x. PMID 17092218
- [Result] Chappuis V, Araujo MG, Buser D. Clinical relevance of dimensional bone and soft tissue alterations post-extraction in esthetic sites. Periodontol 2000. 2017 Feb;73(1):73-83. doi: 10.1111/prd.12167. PMID 28000281
- [Result] Caplanis N, Lozada JL, Kan JY. Extraction defect assessment, classification, and management. J Calif Dent Assoc. 2005 Nov;33(11):853-63. PMID 16463907
- [Result] Perez-Albacete Martinez MA, Perez-Albacete Martinez C, Mate Sanchez De Val JE, Ramos Oltra ML, Fernandez Dominguez M, Calvo Guirado JL. Evaluation of a New Dental Implant Cervical Design in Comparison with a Conventional Design in an Experimental American Foxhound Model. Materials (Basel). 2018 Mar 21;11(4):462. doi: 10.3390/ma11040462. PMID 29561788
- [Result] Li Manni L, Lecloux G, Rompen E, Aouini W, Shapira L, Lambert F. Clinical and radiographic assessment of circular versus triangular cross-section neck Implants in the posterior maxilla: A 1-year randomized controlled trial. Clin Oral Implants Res. 2020 Sep;31(9):814-824. doi: 10.1111/clr.13624. Epub 2020 Jun 29. PMID 32496624
- [Result] Araujo MG, da Silva JCC, de Mendonca AF, Lindhe J. Ridge alterations following grafting of fresh extraction sockets in man. A randomized clinical trial. Clin Oral Implants Res. 2015 Apr;26(4):407-412. doi: 10.1111/clr.12366. Epub 2014 Mar 12. PMID 24621203
- [Result] Belser UC, Grutter L, Vailati F, Bornstein MM, Weber HP, Buser D. Outcome evaluation of early placed maxillary anterior single-tooth implants using objective esthetic criteria: a cross-sectional, retrospective study in 45 patients with a 2- to 4-year follow-up using pink and white esthetic scores. J Periodontol. 2009 Jan;80(1):140-51. doi: 10.1902/jop.2009.080435. PMID 19228100